CLINICAL TRIAL: NCT05640336
Title: Single vs Planned Double-Debridement Antibiotics and Implant Retention Followed by Chronic Antibiotic Suppression for the Treatment of Acute Periprosthetic Joint Infection: A Prospective, Multicenter, Randomized Clinical Trial
Brief Title: Treatment of Acute Periprosthetic Joint Infection Comparing Single and Planned Double-Debridement Antibiotics and Implant Retention Followed by Chronic Antibiotic Suppression
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Columbia University (Other)
Responsible Party: Principal Investigator, Matthew P. Abdel, M.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-006739
Record Dates: First submitted 2022-11-28; First posted 2022-12-07 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Periprosthetic Joint Infection
Keywords: Total knee arthroplasty; Total hip arthroplasty
MeSH Terms: interventions — Debridement; Anti-Bacterial Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single DAIR Surgery Arm (Active Comparator): Subjects will undergo a single Debridement Antibiotics and Implant Retention (DAIR) surgical procedure, along with IV antibiotics and followed by oral suppressive antibiotics. This method is currently used and considered to be standard of care.
  Interventions: Procedure: Single Debridement, Antibiotics and Implant Retention
- Double DAIR Surgery Arm (Active Comparator): Subjects will undergo planned double Debridement Antibiotics and Implant Retention (DAIR) surgical procedure, along with IV antibiotics and followed by oral suppressive antibiotics. This method is currently used and considered to be standard of care.
  Interventions: Procedure: Planned Double Debridement, Antibiotics and Implant Retention

INTERVENTIONS:
Procedure: Single Debridement, Antibiotics and Implant Retention — Surgical debridement and wash out of infected joint. The polyethylene (plastic) insert, which acts as the articulating surface (modular component) of the prosthesis, will be removed and the exposed surfaces scrubbed, sterilized, and soaked. A new modular component will be placed with additional irrigation and antiseptic soak. Tissue cultures will be sent to the lab for further evaluation and antibiotic guidance. After the operation subjects will continue six weeks of IV antibiotics followed by oral antibiotic suppression for the life of the implant or at least two years after operation.
  Arms: Single DAIR Surgery Arm
Procedure: Planned Double Debridement, Antibiotics and Implant Retention — Surgical debridement and wash out of infected joint with an additional irrigation and debridement scheduled for approximately 5 days after the initial DAIR. During the first washout, antibiotic cement beads will be placed in the joint and these will remain in the interim until they are removed during the second washout. During the second DAIR, the antibiotic beads are removed, and the modular components are once again removed and replaced with new components. Exposed surfaces are again irrigated and debrided following a standardized protocol. A six-week course of IV antibiotics will follow the DAIR with additional oral antibiotics for the life of the component (standard of care) or at least a minimum of two years.
  Arms: Double DAIR Surgery Arm

SUMMARY:
The purpose of this research is to evaluate two different standard of care surgeries in treating periprosthetic joint infection (PJI) after total hip and knee arthroplasty. Researchers are looking at differences in outcomes following single versus planned double debridement, antibiotics, and implant retention (DAIR) for acutely infected total hip arthroplasty (THA), and total knee arthroplasties (TKAs).

ELIGIBILITY:
Inclusion Criteria:

* Patients who speak English and are willing to sign the consent form
* Patients with acute early postoperative infection (symptoms ≤ 4 weeks from surgery; symptoms < 4 weeks in duration) and acute hematogenous infection (greater than 4 weeks from surgery; symptoms < 3 weeks in duration) of a primary total knee or total hip arthroplasty, defined as:

  * A sinus communicating with the prosthesis OR
  * Two positive cultures obtained from the prosthesis OR
  * 4 of 5 criteria: Elevated ESR (> 30mm/hr) and CRP (> 10mg/L); Elevated synovial leukocyte count (>3000 cells/μL) or change of ++ on; leukocyte esterase strip; Elevated synovial neutrophil percentage (> 80%); One positive culture; Positive histological analysis of periprosthetic tissue (> 5 neutrophils per high; Power field in 5 high power fields x 400).
* OR Patient with an acute infection diagnosed clinically by an orthopedic surgeon treated with DAIR

Exclusion Criteria:

* Patients with a chronic PJI, defined as: presentation of symptoms > 4 weeks in duration.
* Revision surgery or previous two-stage reimplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Estimated)
Dates: Start 2023-03-03 (Actual); Primary Completion 2032-03 (Estimated); Study Completion 2032-03 (Estimated)

PRIMARY OUTCOMES:
Subjects free from failure | 1 year following DAIR.
  Total number of subjects considered failure free at one year from surgical DAIR procedure. Failure is defined as reoperation for infection within one year from surgical procedure.

SECONDARY OUTCOMES:
Readmission within 90 days of the surgical DAIR procedure | 90 days following DAIR procedure
  Total number of subjects to required hospital readmission within 90 days of DAIR.
1-year surgical reoperation rate | 1 year following DAIR procedure
  Total number of subjects to require reoperation or revision with or without infection within one year from the surgical DAIR procedure.
5-year surgical reoperation rate | 5 years following DAIR procedure
  Total number of subjects to require reoperation or revision with or without infection within five years from the surgical DAIR procedure.
10-year surgical revision rate | 10 years following DAIR procedure
  Total number of subjects to require reoperation or revision with or without infection within ten years from the surgical DAIR procedure.
Hospital length of stay | Approximately 2 weeks following DAIR procedure
  Total number of days subjects were admitted to the hospital
Resource analysis | Approximately 2 weeks following DAIR procedure
  Hospital admission cost comparison between the two study arms
Clinical Outcome Scores | 1, 5, and 10 years following DAIR procedure
  Evaluation of patient reported Harris Hip or Knee Society Scores
Adverse events | 10 years following DAIR procedure
  Total number of subjects to experience adverse events related to either drug or the surgical procedure
Survivorship | 10 years following DAIR procedure
  Total number of subject deaths post-surgical DAIR procedure

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Abdel, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic Florida, Jacksonville, Florida
  - Mayo Clinic Minnesota, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials